CLINICAL TRIAL: NCT06588075
Title: Evaluation of the Accuracy of Zygomatico-Maxillary Complex Fracture Reduction and Fixation Using a Full Digital Workflow Versus Conventional Protocol: a Randomized Clinical Trial
Brief Title: A Full Digital VS Conventional Protocol in Management of Zygomatico-Maxillary Complex Fracture
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Ayman Fayek, Assistant lecturer in Oral and Maxillofacial department in Future university in Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMFS 3319
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Zygomatic Fractures
Keywords: Zygomatic fracture; computer guided surgery; patient specific implant; predictive holes surgical guide; Zygomatico-Maxillary complex fracture
MeSH Terms: conditions — Zygomatic Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental): all cases that will be allocated in this group will undergo treatment using a full digital protocol depending on planning software and the planning will be carried out into the operating room using 3D printed predictive holes surgical guides to determine accurately the optimum position of customized plates
  Interventions: Procedure: Reduction and fixation of zygomatico- Maxillary complex fracture using a full digital work flow
- control group (Active Comparator): patients in this group will be treated using a conventional protocol of reduction depending on visualization intraoperative and tactile sensation and will be fixed using a stock miniplates and screws.
  Interventions: Procedure: Reduction and fixation of zygomatico- maxillary complex fracture using a conventional free hand protocol

INTERVENTIONS:
Procedure: Reduction and fixation of zygomatico- Maxillary complex fracture using a full digital work flow — All surgeries will be carried out under general anesthesia the fracture lines will be exposed then For the study group: following the exposure of all fracture lines , anatomically seated bone-supported predictive holes surgical guides will be inserted on the bone segments with intimate contact. Each segment hole will be drilled according to the predesigned predictive holes guide. The fractured segments will then be reduced and fixed using titanium miniplates customized for the patient and screws at least two screws for each fracture segment. then closure in layers will be performed using absorbable vicryl for deep layers and intraoral sutures and non-absorbable polyproline for skin closure.
  Arms: study group
Procedure: Reduction and fixation of zygomatico- maxillary complex fracture using a conventional free hand protocol — For the control group: all cases will be treated under general anesthesia and the fracture lines will be exposed then the conventional protocol of treatment depend mainly on visualization of the fracture line and tactile sensation of the operator intra-operative during reduction procedure and the fixation of fractured segments will be done using titanium miniplates and screws then closure in layers will be performed.
  Arms: control group

SUMMARY:
this study aims To evaluate The Accuracy of Zygomatico- Maxillary Complex (ZMC) Fracture reduction and fixation Using customized Patient-Specific implant and patient-specific predictive holes surgical guide Versus Conventional Technique of reduction and fixation.

DETAILED DESCRIPTION:
The ZMC has multiple points of articulation with the craniofacial skeleton making accurate assessment of reduction at all articulations intraoperative in multiple planes very challenging and the interference of soft tissue edema and a narrowed visual field increases the possibility of intraoperative overcorrection or underestimation of pre-injured position of all fracture lines at the same time resulting in a suboptimal reduction. As a trial to maximize the benefits of digital planning carrying the plan into a real operating room using a patient-specific surgical guide to predrill screw holes and guide patient-specific implants during fixation according to the planning depend on CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Zygomatic Fracture Types III, IV, V, VII, and VIII according to Rowe and Killey's classification.
* Age range (18-60 years).
* Patients are willing for the surgical procedure and follow-up, with informed consent

Exclusion Criteria:

* Zygomatic Fracture Type I, II according to Rowe and Killey's classification.
* Patients with contraindications for general anesthesia.
* Patient on radiotherapy.
* Patients suffer from bone disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Zygomatic reposition | immediate postoperative
  the accuracy of zygomatic bone reduction and fixation using postoperative CT scan

SECONDARY OUTCOMES:
intraoperative time | during the operation
  duration of operation using stopwatch
paresthesia | pre operative, immediate postoperative and 6 months post operative
  sensation in the area supplied by the infraorbital nerve using a 2 points discrimination test
patient satisfaction | 6 months postoperative
  patient aesthetic satisfaction will be measured using a visual analogue scale from 0 to 10 in a questionnaire form, zero mean not satisfied at all and 10 is the maximum satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Ayman Fayek, M.Sc, Principal Investigator — Assistant lecturer oral and maxillofacial surgery department Future university in Egypt
Locations (1):
- Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
the data will be available from the corresponding author upon reasonable request.